CLINICAL TRIAL: NCT03950713
Title: Taiwanese Mindfulness Program for Long Term Residents With Type 2 Diabetes
Brief Title: Mindfulness Program for Older-Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FYH-IRB-1040602
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2016-08

CONDITIONS: Mental Health Wellness 1
Keywords: Mindfulness-based Program; Relocation stress; Depression; Glycemic control
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial was used to examine the effectiveness of the MBSR-T. The outcomes included HbA1c levels progression as the primary endpoint, and relocation stress, depression as secondary end points. Participants in the intervention group received the MBSR-T in addition to routine care. The control group received the routine care provided in facilities, including routine check-ups at diabetes clinics as necessary.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction Program - Taiwan (MBSR-T) (Experimental): Participants in the intervention group received the MBSR-T in addition to routine care.
  Interventions: Behavioral: Mindfulness-based Stress Reduction Program - Taiwan (MBSR-T)
- Routine care (No Intervention): The control group received the routine care provided in facilities, including routine check-ups at diabetes clinics as necessary.

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction Program - Taiwan (MBSR-T) — The MBSR-T is focused on strategies to manage diabetes distress for new residents by three new techniques. Firstly, it involves practicing body and meditation exercises for openness to the awareness and acceptance of transferred life experiences, such as mindful attention exercise, which is assumed to allow the residents to behave in a less reactive and more reflective manner when confronted with transferred life stressors. Second, mindfulness meditation techniques were provided for difficult thoughts and feelings related to diabetes, such as paying full attention to the present moment of life and choosing to respond skillfully rather than reacting automatically to external events, thoughts or emotions as they arise. Third, a specific topic, for example on how to be mindful when life style is changed, or how to pay attention to the present moment within Chinese culture of peacefulness was discussed in each session.
  Arms: Mindfulness-based Stress Reduction Program - Taiwan (MBSR-T)

SUMMARY:
This study aimed to evaluate the effectiveness of the newly developed Mindfulness-Based Stress Reduction-Taiwan program (MBSR-T) for old people with type 2 diabetes living in long-term care facilities.

DETAILED DESCRIPTION:
This study reported the first randomized controlled trial of Mindfulness-based reduction stress for residents with type 2 diabetes newly moved into long-term care facilities on depression, relocation stress and HbA1c levels. The results highlighted the benefits of using strategies in the MBSR-T to promote good quality of diabetes care for residents in long-term care.

The contents of the 9-week MBSR-T program were adapted from an initial MBSR program by the Taiwan Mindfulness Association for older people with diabetes (Chinese version). The program consisted of a 1.5-hour session each week for 9-weeks for a group of 8 to 10 participants. Each session included 30 minutes of mindful deep breathing relaxation and 60 minutes of practicing mindfulness activities.

A total sample of 140 was determined. All eligible individuals in each long-term care facility were randomized by computerized random numbers, sequence generated by an independent statistician with one-to-one ratio for allocating to either control or intervention group. All participants were blinded to group allocation. Participants in the control group received usual care, while participants in the intervention group received the MBSR-T in addition to the usual care. All sessions in the MBSR-T were delivered by a trained mindfulness registered nurse who had received additional trainer qualification of mindfulness. A research assistant was blinded to the study protocol, who was employed to undertake data collection at baseline, at 3, 6, and 9 weeks (T0, T1, T2, T3).

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85 years old
* Diagnosed with type 2 diabetes
* Moving into the facility within a year
* No obvious delirium, confusion or current psychiatric illness
* Being able to communicate in Chinese.

Exclusion Criteria:

* Terminally ill
* Unable to communicate in Chinese.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
HbA1c values | Change from baseline HbA1c values at 12 weeks
  Glycemic control was measured by HbA1c values, and data were collected from participants' medical records.

SECONDARY OUTCOMES:
Relocation Stress Scale | Change from baseline relocation stress mean scores at 9 weeks
  Relocation Stress Scale (Chinese version), This scale is a 29-item functional assessment of health status with a 5-point Likert scale (5 is the highest relocation stress, 1 is the lowest). The internal consistency .72 has been reported.
Depression and Anxiety Stress Scale (DASS-21) | Change from baseline depression and anxiety stress mean scores at 9 weeks
  The Depression and Anxiety Stress Scale (DASS-21) was used to measure depression. The DASS-21 in Chinese version consists of 21 items with a 4-point Likert scale. The good internal consistency for the DASS-21 subscales .92 for depression, .94 for anxiety, and .91 for stress have been reported.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Ming Chen, Study Chair — Fooyin University
Locations (1):
- Fooyin University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
In the study consent form, the participants only singe their agreements for this study authors, not for other researchers.